CLINICAL TRIAL: NCT06018441
Title: National, Multicenter, Non-interventional, Prospective Study to Explore the Quality of Life of Patients With Severe Asthma Starting Treatment With Dupilumab (Dupixent®) in a Real-world Setting
Brief Title: A Study to Evaluate the Quality of Life in Male and Female Adult Participants With Severe Asthma Treated With Dupilumab in a Real-world Setting
Acronym: PROVERB
Status: Completed | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: OBS17526; U1111-1279-3274 (Registry Identifier: ICTRP)
Record Dates: First submitted 2023-08-24; First posted 2023-08-30 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Severe asthma: Participants with severe asthma starting treatment with dupilumab

SUMMARY:
Primary Objective:

- To describe dupilumab health-related quality of life (HRQoL) effectiveness at 52 weeks compared to baseline.

Secondary Objectives:

* To describe dupilumab HRQoL effectiveness at 12 and 24 weeks compared to baseline.
* To assess the safety during the year of treatment in a real-world setting.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be at least 18 years of age inclusive, at the time of signing the informed consent.
* Participant for whom decision of initiation and prescription of dupilumab (Dupixent®) for the severe uncontrolled asthma indication was made by the investigator within four weeks before the inclusion in the study. Oral CorticoSteroid (OCS) or non-OCS-dependent patient could be included.
* Participant for whom St. George's Respiratory Questionnaire (SGRQ) score is available within the last 4 weeks prior to dupilumab initiation. SGRQ score could be collected at baseline visit for participants who have not yet started dupilumab.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

* Participant below 18 years of age. - Participant participating in a clinical trial at the time of enrolment.
* Participant under guardianship, trusteeship or under judicial protection.

The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with severe asthma
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2023-10-03 (Actual); Primary Completion 2025-10-10 (Actual); Study Completion 2025-10-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in health-related quality of life (HRQoL), as measured by the St. George's Respiratory Questionnaire (SGRQ) | Baseline (Day 0), Week 52
  The SGRQ is a 50-item questionnaire designed to measure and quantify health status in adult participants with chronic airflow limitation. A global score ranges from 0 to 100. Scores by dimension are calculated for 3 domains: Symptoms, Activity and Impacts (Psycho-social) as well as a total score. A lower score indicates better quality of life.

SECONDARY OUTCOMES:
Change from baseline in health-related quality of life (HRQoL), as measured by the St. George's Respiratory Questionnaire (SGRQ) | Baseline (Day 0), Week 12 and Week 24
  The SGRQ is a 50-item questionnaire designed to measure and quantify health status in adult participants with chronic airflow limitation. A global score ranges from 0 to 100. Scores by dimension are calculated for 3 domains: Symptoms, Activity and Impacts (Psycho-social) as well as a total score. A lower score indicates better quality of life.
Number of participants with adverse events (AEs) | Day 0 to Week 52
Number of participants with serious adverse events (SAEs) | Day 0 to Week 52
Number of participants with adverse events of special interest | Day 0 to Week 52
Number of participants with medication errors | Day 0 to Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site, France, France

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org